CLINICAL TRIAL: NCT03120364
Title: A Randomized, Double Blinded, Multi-center Phase III Confirmatory Study to Assess the Immunogenicity and Safety of NBP608 Compared to Zostavax in Healthy Adult Aged 50 and Over
Brief Title: Immunogenicity and Safety of NBP608 Compared to Zostavax in Healthy Adult Aged 50 and Over
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NBP608_HZ_III_2015
Record Dates: First submitted 2017-04-12; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Herpes Zoster
Keywords: Herpes Zoster Vaccine; Prevention of Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBP608 (Experimental): Single dose 0.5mL of NBP608 by subcutaneous injection into the outer aspect of the upper arm
  Interventions: Biological: NBP608
- Zostavax (Active Comparator): Single dose 0.65mL of Zostavax by subcutaneous injection into the outer aspect of the upper arm
  Interventions: Biological: Zostavax

INTERVENTIONS:
Biological: NBP608 — Preparation of Oka/SK strain of live, attenuated zoster virus
  Arms: NBP608
Biological: Zostavax — Preparation of Oka/Merck strain of live, attenuated zoster virus
  Arms: Zostavax

SUMMARY:
This study assesses non-inferiority by comparing GMR(Geometric Mean Ratio) of NBP608 to Zostavax which are evaluated by gpELISA (Glycoprotein Enzyme Linked Immunosorbent Assay). Total of 824 healthy subjects (412 subjects per treatment arm) aged 50 and over are enrolled, and each subject is administered with single dose of vaccine which is randomly assigned.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double blinded, parallel-group study to assess the Immunogenicity and safety of NBP608 compared to Zostavax which are indicated for the prevention of herpes zoster. Total of 824 healthy subjects aged 50 and over are enrolled, and each subject is administered with single dose of vaccine which is randomly assigned in 1:1 ratio. Stratified randomization for age group is used to achieve the balance of treatment assignment within age strata.

Total of five visits are scheduled including two visits via telephone contact. Blood sampling is conducted for immunogenicity assessment before and 6 weeks after vaccination at Visit 2 and Visit 4 respectively. Safety is monitored 1 week, 6 weeks and 26 weeks after vaccination through Visit 3*, Visit 4 and Visit 5* (* telephone contact)

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult over aged 50 years
* Menopause females or females who are confirmed to be negative in a preganacy test on the day of screening and agree to practice birth control for 6 weeks after signing informed concent

Exclusion Criteria:

* Those with hypersensitivity to any component of IP(Investigational Product), such as gelatin
* Those with a history of hypersensitivity to vaccination, such as Guillain-Barre syndrome
* Those who have received antiviral agents witin 1 month prior to IP vaccination (topical antiviral agent is allowed)
* Those who have previously received herpes zoster vaccine
* Those who have a history of herpes zoster
* Those with congenital or acquired immunodeficiency
* Those with active untreated tuberculosis
* Those who have received blood products or immunoglobulin within 3 months prior to IP(Investigational Products) vaccination
* Those who have received other IPs(Investigational Products) in another clinical study witin 4 weeks prior to IP vaccination in this study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 824 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2015-12-16 (Actual); Study Completion 2016-04-28 (Actual)

PRIMARY OUTCOMES:
GMR(Geometric Mean Ratio) of VZV(Varicella-Zoster Virus) antibody titer measured by gpELISA(Glycoprotein Enzyme-Linked Immnosorbent Assay) | 6 weeks after IP(Investigational Product) vaccination
  The geometric mean fold rise of subjects' VZV(Varicella zoster virus) antibody titers of NBP608 from prevaccination to 6weeks postvaccination
GMR(Geometric Mean Ratio) ratio of NBP608 to Zostavax measured by gpELISA | 6 weeks after IP(Investigational Product) vaccination
  Non-inferiority assessment by comparing GMR(Geometric Mean Ratio) of NBP608 to Zostavax

SECONDARY OUTCOMES:
VZV-CMI(Varicella Zoster Virus-Cell Mediated Immnogenicity) response measured by IFN-γ(Interferon-gamma) ELISPOT (Enzyme-Linked Immunospot) | 6 weeks after IP(Investigational Product) vaccination
VZV-CMI(Varicella Zoster Virus-Cell Mediated Immnogenicity) response measured by IL-2(Interleukin-2) ELISPOT (Enzyme-Linked Immunospot) | 6 weeks after IP(Investigational Product) vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Jin Cheong, Ph.D, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, Guro-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Oliveira Gomes J, Gagliardi AM, Andriolo BN, Torloni MR, Andriolo RB, Puga MEDS, Canteiro Cruz E. Vaccines for preventing herpes zoster in older adults. Cochrane Database Syst Rev. 2023 Oct 2;10(10):CD008858. doi: 10.1002/14651858.CD008858.pub5. PMID 37781954
- [Derived] Choi WS, Choi JH, Jung DS, Choi HJ, Kim YS, Lee J, Jang HC, Shin EC, Park JS, Kim H, Cheong HJ. Immunogenicity and safety of a new live attenuated herpes zoster vaccine (NBP608) compared to Zostavax(R) in healthy adults aged 50 years and older. Vaccine. 2019 Jun 12;37(27):3605-3610. doi: 10.1016/j.vaccine.2019.04.046. Epub 2019 May 20. PMID 31122860